CLINICAL TRIAL: NCT01207921
Title: A Pilot Study of Lenalidomide Maintenance Therapy Following Autologous Stem Cell Transplantation in Patients With Relapsed/Refractory Hodgkin Lymphoma
Brief Title: Lenalidomide Maintenance Therapy Post Autologous Transplant for Hodgkins Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201010719
Record Dates: First submitted 2010-09-21; First posted 2010-09-23 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Hodgkin Disease
MeSH Terms: conditions — Hodgkin Disease | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): Lenalidomide 15 mg/day Cycle 1 (28 days).
  If no unacceptable side effects Cycle 2 (28 days) will be lenalidomide 20 mg/day.
  If no unacceptable side effects Cycles 3 thru 18 (28 days for each cycle) will be lenalidomide 25 mg/day.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide
  Other Names: Revlimid

SUMMARY:
The purpose of this study to evaluate the feasibility of lenalidomide maintenance therapy in patients with relapsed Hodgkin lymphoma after autologous transplant

DETAILED DESCRIPTION:
Primary Objectives

-To evaluate the feasibility of lenalidomide maintenance therapy in patients with relapsed Hodgkin lymphoma after autologous stem cell transplant, as measured by dropout rate.

Secondary Objectives

* To assess overall survival, event free survival, and progression free survival.
* To establish the adverse event profile of long-term maintenance therapy with lenalidomide in this patient population.
* To assess the conversion of partial response/stable disease post-ASCT to complete response.
* To evaluate changes in immune cell number and function and plasma proteins before, during, and after lenalidomide therapy (correlative studies).

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically documented classical Hodgkin lymphoma that is recurrent or refractory to standard chemotherapy.
* Core biopsies are acceptable if they contain adequate tissue for primary diagnosis and immunophenotyping. If the original diagnostic specimen is not available, relapsed or refractory specimens may be used. Bone marrow biopsies as the sole means of diagnosis are not acceptable; however, they may be used in conjunction with nodal biopsies. Fine needle aspirates (FNA) are not acceptable. Pathology reports must be submitted with the appropriate CRFs, and the actual biopsy specimens are not requested for central review. Patients with cHL have one of the following WHO subtypes:

  * Nodular sclerosis Hodgkin lymphoma
  * Lymphocyte-rich Hodgkin lymphoma
  * Mixed cellularity Hodgkin lymphoma
  * Lymphocyte-deplete Hodgkin lymphoma cHL patients without one of these subtypes designated cHL not otherwise specified are also eligible.

NOTE: Patients with nodular lymphocyte-predominant HL are not eligible.

* Patient must have undergone autologous stem cell transplant (ASCT) between 60 and 90 days prior to study registration.
* Patient must be ≥ 18 years old.
* Patient must have an ECOG performance status of ≤ 2 at study entry.
* Patient must have adequate hematologic, renal, and hepatic function as defined by:

  * Absolute neutrophil count ≥ 1000 / μL
  * Platelets ≥ 30,000 / μL
  * Serum creatinine ≤ 1.5 X institution upper limit of normal (ULN)
  * Total bilirubin ≤ 1.5 mg/dL
  * AST (SGOT) and ALT (SGPT) ≤ 3 x ULN (if not attributed to cHL)
* Patient must be disease free of prior malignancies for ≥ 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
* Patient must understand and voluntarily sign an informed consent form.
* Patient must be able to adhere to the study visit schedule and other protocol requirements.
* If a female of childbearing potential (FCBP), patient must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) for at least 28 days before starting study drug; 2) while participating in the study; and 3) for at least 28 days after discontinuation from the study. The two methods of reliable contraception must include one highly effective method (i.e. intrauterine device (IUD), hormonal [birth control pills, injections, or implants], tubal ligation, partner's vasectomy) and one additional effective (barrier) method (i.e. latex condom, diaphragm, cervical cap). FCBP must be referred to a qualified provider of contraceptive methods if needed
* A FCBP is defined as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* A FCBP must have two negative pregnancy tests (sensitivity of at least 50 mIU/mL) prior to starting study drug. The first pregnancy test must be performed within 10-14 days prior to the start of study drug and the second pregnancy test must be performed within 24 hours prior to prescribing the study drug. The subject may not receive study drug until the Investigator has verified that the results of these pregnancy tests are negative.
* If male, patient must agree to use a latex condom during sexual contact with FCBP while participating in the study and for at least 28 days following discontinuation from the study even if he has undergone a successful vasectomy.
* Patient must be able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).
* Patient must be registered into the mandatory Revlimid REMS® program and be willing and able to comply with the requirements of Revlimid REMS®.

Exclusion Criteria:

* Patient who has undergone allogeneic stem cell transplantation.
* Patient who shows evidence of progressive disease during salvage chemotherapy or following ASCT.
* Patient has any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent him/her from signing the informed consent form.
* Patient has any condition, including the presence of laboratory abnormalities, which places him/her at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Patient has used any other anti-cancer drug or therapy, including experimental, within 30 days of initiation of lenalidomide treatment (radiation therapy is allowed within 30 days).
* Patient has known hypersensitivity to thalidomide.
* Patient developed erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Patient has any prior use of lenalidomide.
* Patient is known to be positive for HIV or infectious hepatitis, type A, B, or C.
* Patient is pregnant or breastfeeding.
* Patient has concurrent use of other anti-cancer agents or treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-04-28 (Actual); Primary Completion 2016-09-19 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility of lenalidomide maintenance therapy in patients with relapsed Hodgkin lymphoma after ASCT, as measured by dropout rate. | 12 months
  Will be described by the proportion of patients who drop out of the study for drug-related reasons at or before 12 months

SECONDARY OUTCOMES:
Overall survival (OS) | Until death (estimated to be 10 years)
Adverse event profile | From start of treatment through 30 days following completion of treatment
  To establish the adverse event profile of long-term maintenance therapy with lenalidomide in this patient population.
Conversion of partial response/stable disease post-ASCT to complete response. | 1 year
  To assess the conversion of partial response/stable disease post-autologous stem cell transplant to complete response.
Evaluate immune response | Through 30 days after end of treatment
  To evaluate changes in immune cell number and function and plasma proteins before, during, and after lenalidomide therapy (correlative studies).
Event-free survival (EFS) | Until progression or death (whichever comes first) - estimated to be 10 years
Progression-free survival (PFS) | Until progression (estimated to be 10 years)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Fehniger, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - Washington University School of Medicine, St Louis, Missouri
  - Wake Forest University, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartlett NL. Modern treatment of Hodgkin lymphoma. Curr Opin Hematol. 2008 Jul;15(4):408-14. doi: 10.1097/MOH.0b013e328302c9d8. PMID 18536581
- [Background] Fehniger, T.A., et al., A Phase II Multicenter Study of Lenalidomide in Relapsed or Refractory Classical Hodgkin Lymphoma. ASH Annual Meeting Abstracts, 2009. 114(22): p. 3693-.
- [Background] Boll B, Borchmann P, Topp MS, Hanel M, Reiners KS, Engert A, Naumann R. Lenalidomide in patients with refractory or multiple relapsed Hodgkin lymphoma. Br J Haematol. 2010 Feb;148(3):480-2. doi: 10.1111/j.1365-2141.2009.07963.x. Epub 2009 Oct 15. No abstract available. PMID 19863533
- [Background] Attal, M., et al., Lenalidomide After Autologous Transplantation for Myeloma: First Analysis of a Prospective, Randomized Study of the Intergroupe Francophone Du Myelome (IFM 2005 02). ASH Annual Meeting Abstracts, 2009. 114(22): p. 529-.
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu